CLINICAL TRIAL: NCT07254988
Title: Gut Peptides and Bone Remodeling in Children With Neuromuscular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bolette Hartmann, Principal investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TK-23
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Spinal Muscular Atrophy (SMA); Cerebral Palsy (CP); Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Atrophy, Spinal; Cerebral Palsy; Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal test (Experimental): Oral liquid meal test
  Interventions: Other: Meal test
- Glucose dependent insulinotropic polypeptide (GIP) + Glucagon-like-peptide 2 (GLP-2) (Experimental): Subcutaneous co-injection of GIP and GLP-2
  Interventions: Other: GIP + GLP-2
- Placebo (Placebo Comparator): Subcutaneous injection of saline
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Meal test — Ingestion of an oral liquid meal (nutridrink), 3.3 mL/kg body weight.
  Arms: Meal test
Other: GIP + GLP-2 — Subcutaneous GIP + GLP-2 injection (1 mL containing 100 microgram GIP + 1 mL containing 400 microgram GLP-2).
  Arms: Glucose dependent insulinotropic polypeptide (GIP) + Glucagon-like-peptide 2 (GLP-2)
Other: Placebo — Subcutaneous saline injection (2 mL isotonic saline).
  Arms: Placebo

SUMMARY:
Both GIP and GLP-2 reduce bone resorption (measured as CTX) in healthy adult individuals. In this study, we will investigate whether GIP and GLP-2 reduce CTX in children with spinal muscular atrophy, duchenne muscular dystrophy, or cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis with Cerebral palsy (CP), Duchenne muscular dystrophy (DMD) or Spinal muscular atrophy (SMA) resulting in the need of a wheelchair

Exclusion Criteria:

* Use of anti-resorptive medication
* Confounding illnesses
* Pregnancy
* Allergy towards the components given on the test days
* Hgb<6.5 mmol/L

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CTX | -10 to 240 minutes
  Bone resorption measured as carboxy-terminal telopeptide of type I collagen (CTX)

SECONDARY OUTCOMES:
P1NP | -10 to 240 minutes
  Bone formation measured as procollagen type I N-terminal propeptide (P1NP)
PTH | -10 to 240 minutes
  Parathyroid hormone (PTH) measured in plasma
Glucose | -10 to 240 minutes
  Blood glucose measured in plasma
GIP | -10 to 240 minutes
  Glucose-dependent insulinotropic polypeptide (GIP) measured in plasma
GLP-2 | -10 to 240 minutes
  Glucagon-like-peptide 2 (GLP-2) measured in plasma
Blood pressure | -10 to 240 minutes
  Measured before blood sampling
Heart rate | -10 to 240 minutes
  Measured before blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Mette Marie Rosenkilde, Study Director — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No